CLINICAL TRIAL: NCT07227454
Title: A Double-blind, Randomized, Psychoactive Placebo-controlled Study to Evaluate the Efficacy and Safety of Intranasal Esketamine 84 mg in Addition to Comprehensive Standard of Care for the Rapid Reduction of the Symptoms of Major Depressive Disorder in Adolescent Participants With Acute Suicidal Ideation or Behavior
Brief Title: A Study to Evaluate the Efficacy and Safety of Esketamine for Reduction of Symptoms of Major Depressive Disorder
Acronym: AVENUE
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 54135419SUI3003; 54135419SUI3003 (Other: Janssen Research & Development, LLC); 2024-518615-19-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2025-11-11; First posted 2025-11-12 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Esketamine; Midazolam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Intranasal Esketamine + Oral Placebo (Experimental): Participants will receive intranasal esketamine 84 milligrams (mg) along with oral placebo solution twice weekly for 4 weeks (Days 1, 4, 8, 11, 15, 18, 22, and 25). On Day 4 a decrease to intranasal esketamine 56 mg (in a blinded fashion per investigator's judgment) is permitted. Thereafter, dose may be flexed between 56 mg and 84 mg during the treatment period.
  Interventions: Drug: Esketamine; Other: Oral Placebo
- Intranasal Placebo + Oral Midazolam (Placebo Comparator): Participants will receive oral midazolam (0.0625 milligrams per kilograms [mg/kg]) and intranasal placebo twice weekly for 4 weeks (Days 1, 4, 8, 11, 15, 18, 22, and 25). On Day 4 a sham decrease to esketamine 56 mg dose (in a blinded fashion per investigator's judgment) is permitted. Thereafter, sham dose may be flexed between 56 mg and 84 mg during the treatment period.
  Interventions: Drug: Midazolam; Other: Intranasal Placebo

INTERVENTIONS:
Drug: Esketamine — Esketamine will be administered as intranasal solution.
  Other Names: JNJ-54135419
  Arms: Intranasal Esketamine + Oral Placebo
Drug: Midazolam — Midazolam will be administered as oral solution.
  Arms: Intranasal Placebo + Oral Midazolam
Other: Oral Placebo — Placebo will be administered as oral solution.
  Arms: Intranasal Esketamine + Oral Placebo
Other: Intranasal Placebo — Intranasal placebo will be administered as nasal solution.
  Arms: Intranasal Placebo + Oral Midazolam

SUMMARY:
The purpose of this study is to evaluate how well JNJ-54135419 works (efficacy) in addition to comprehensive standard of care (SoC) in rapidly reducing the symptoms of major depressive disorder (MDD, a mental disorder characterized by a persistent feeling of sadness and loss of interest in activities) as compared with psychoactive placebo (does not contain JNJ-54135419) plus SoC in adolescent participants with acute suicidal ideation or behavior.

ELIGIBILITY:
Inclusion Criteria:

* Must meet diagnostic and statistical manual of mental disorders (5th edition) (DSM-5) diagnostic criteria for major depressive disorder (MDD) based upon clinical assessment and confirmed by the mini-international neuropsychiatric interview for children and adolescents (MINI-KID)
* Must have a clinical global impression - severity of suicidality - revised (CGI-SS-R) score of "Markedly" or greater (that is, greater than or equal to [>=] 4) at both screening and baseline (predose) visits
* Must have a children's depression rating scale - revised (CDRS-R) total score >= 58 at baseline (predose)
* In the physician's opinion, acute psychiatric hospitalization is clinically warranted due to subject's acute suicidality
* Must be medically stable based on physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening

Exclusion Criteria:

* Participant has a current DSM-5 diagnosis of bipolar (or related disorders), intellectual disability, autism spectrum disorder, conduct disorder, oppositional defiant disorder
* Participant currently meets DSM-5 criteria for borderline personality disorder
* Participant has a current or prior DSM-5 diagnosis of a psychotic disorder, or MDD with psychosis
* Participant has a history of seizure disorder
* Participant has known allergies, hypersensitivity, intolerance or contraindications to midazolam, esketamine or ketamine, or their excipients

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 258 (Estimated)
Dates: Start 2026-01-08 (Actual); Primary Completion 2031-04-09 (Estimated); Study Completion 2031-09-15 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Depressive Symptoms Measured by Children's Depression Rating Scale - Revised (CDRS-R) Total Score at 24 Hours Post First Dose | Baseline (pre-dose on Day 1) and 24 hours post first dose (i.e., Day 2)
  The CDRS-R is a 17-item, clinician-reported outcome measure of children's depressive symptom severity. Out of the 17-item, 3 items were non-verbal behavior (listless speech, hypoactivity, and depressed affect) rated on a 5 point scale from 1 (no depression) to 5 (severe depression) and 14 items were rated on a 7-point scale from 1 (no depression) to 7 (severe depression), where higher score indicated more severe depression. The CDRS-R total score was the sum of the 17-tems score and it ranged from 17 (normal) to 113 (severe depression). Higher score indicated more severe depression and worse outcome.

SECONDARY OUTCOMES:
Change from Baseline in CDRS-R Total Score at Day 25 | Baseline (predose on Day 1) and Day 25 (4 hours post dose)
  The CDRS-R is a 17-item, clinician-reported outcome measure of children's depressive symptom severity. Out of the 17-item, 3 items were non-verbal behavior (listless speech, hypoactivity, and depressed affect) rated on a 5-point scale from 1 (no depression) to 5 (severe depression) and 14 items were rated on a 7-point scale from 1 (no depression) to 7 (severe depression), where higher score indicated more severe depression. The CDRS-R total score was the sum of the 17-tems score and it ranged from 17 (normal) to 113 (severe depression). Higher score indicated more severe depression and worse outcome.
Change from Baseline in Clinical Global Impression - Severity of Suicidality - Revised (CGI-SS-R) Score at 24 Hours Post First Dose | Baseline (pre-dose on Day 1) and 24 hours post first dose (i.e., Day 2)
  The CGI-SS-R is a single item clinician-rated measure of the severity of participants' suicidality. The CGI-SS-R asks clinicians to rate the severity of a participant's suicidality using a 7-point scale that ranges from 0 (normal, not at all suicidal) to 6 (among the most extremely suicidal patients). Higher scores indicate greater severity.
Change From Baseline in Symptoms of MDD During the Double-Blind (DB) Treatment Phase as Measured by CDRS-R Total Score | From Baseline up to Day 25
  The CDRS-R is a 17-item, clinician-reported outcome measure of children's depressive symptom severity. Out of the 17-item, 3 items were non-verbal behavior (listless speech, hypoactivity, and depressed affect) rated on a 5-point scale from 1 (no depression) to 5 (severe depression) and 14 items were rated on a 7-point scale from 1 (no depression) to 7 (severe depression), where higher score indicated more severe depression. The CDRS-R total score was the sum of the 17-tems score and it ranged from 17 (normal) to 113 (severe depression). Higher score indicated more severe depression and worse outcome.
Percentage of Participants with Remission of Depressive Symptoms During the DB Treatment Phase | Up to Day 25
  Remission of depressive symptoms is defined as a CDRS-R total score of both less than or equal to (<=) 28 and <= 34 during the DB treatment phase. The CDRS-R is a 17-item, clinician-reported outcome measure of children's depressive symptom severity. Out of the 17-item, 3 items were non-verbal behavior (listless speech, hypoactivity, and depressed affect) rated on a 5 point scale from 1 (no depression) to 5 (severe depression) and 14 items were rated on a 7-point scale from 1 (no depression) to 7 (severe depression), where higher score indicated more severe depression. The CDRS-R total score was the sum of the 17-tems score and it ranged from 17 (normal) to 113 (severe depression). Higher score indicated more severe depression and worse outcome.
Percentage of Responders on Depressive Symptoms During the DB Treatment Phase | Up to Day 25
  Responders on depressive symptoms is defined as >= 50 percent (%) improvement in CDRS-R total score from baseline during the DB treatment phase. The CDRS-R is a 17-item, clinician-reported outcome measure of children's depressive symptom severity. Out of the 17-item, 3 items were non-verbal behavior (listless speech, hypoactivity, and depressed affect) rated on a 5 point scale from 1 (no depression) to 5 (severe depression) and 14 items were rated on a 7-point scale from 1 (no depression) to 7 (severe depression), where higher score indicated more severe depression. The CDRS-R total score was the sum of the 17-tems score and it ranged from 17 (normal) to 113 (severe depression). Higher score indicated more severe depression and worse outcome.
Percentage of Participants with Resolution of Suicidality During the DB Treatment Phase | Up to Day 25
  Participants with resolution of suicidality is defined as a score of 0 (normal, not at all suicidal) or 1 (questionably suicidal) on CGI SS-R, during the DB treatment phase. The CGI-SS-R asks clinicians to rate the severity of a participant's suicidality using a 7-point scale that ranges from 0 (normal, not at all suicidal) to 6 (among the most extremely suicidal patients). Higher score indicate greater severity.
Change From Baseline in Severity of Suicidality As Measured by Clinical Global Impression - Severity of Suicidality - Revised (CGI-SS-R) During the DB Treatment Phase | From Baseline up to Day 25
  The CGI-SS-R is a single item clinician-rated measure of the severity of participants' suicidality. The CGI-SS-R asks clinicians to rate the severity of a participant's suicidality using a 7-point scale that ranges from 0 (normal, not at all suicidal) to 6 (among the most extremely suicidal patients). Higher score indicate greater severity.
Change From Baseline in Clinician-Reported Frequency of Suicidal Thinking (FoST-ClinRO) During the DB Treatment Phase | From Baseline up to Day 25
  FoST-ClinRO is a clinician-rated measure used to assess a participant's frequency of suicidal thinking assessed during the DB treatment phase. The measure uses a 6-point Likert scale that ranges from 0=Never, to 5=All of the time to assess suicidal thinking frequency, where higher scores indicate a more severe condition.
Change from baseline in Patient-Reported Frequency of Suicidal Thinking (FoST-PRO) During the DB Treatment Phase | From Baseline up to Day 25
  FoST-PRO is a single item participant reported measure of the frequency of one's suicidal thinking right now. The single item asks participants to rate the frequency with which they have suicidal thoughts (0 = I have no suicidal thoughts, 1 = I have suicidal thoughts a little of the time, 2 = I have suicidal thoughts some of the time, 3 = I have suicidal thoughts most of the time, and 4 = I have suicidal thoughts all of the time). Higher scores indicate greater severity.
Change from Baseline in Patient Health Questionnaire, 9-item Modified for Adolescents (PHQ-A) Total Score During the DB Treatment Phase | From Baseline up to Day 25
  The PHQ-A is a modified version of the PHQ-9 scale, specifically designed to measure depressive symptom severity in adolescents. A 10-item version of the PHQ-A will be used in this study; the first 9 items assess depressive symptoms. Adolescents use a 4 point Likert scale to rate the severity of their symptoms over the past 2 weeks (range: 0 = not at all to 3 = nearly every day). The PHQ-A total score is the sum of all item responses. The total score can be used to classify adolescents based on the severity of their depressive symptoms: 0-4 (no or minimal depression), 5-9 (mild depression), 10-14 (moderate depression), 15-19 (moderately severe depression), and 20-27 (severe depression). The tenth PHQ-A item measures the degree to which adolescents experience functional difficulties due to their depressive symptoms. Higher scores indicate greater depressive symptoms.
Change From Baseline in KIDSCREEN-10 Total Score During the DB Treatment Phase | From Baseline up to Day 25
  KIDSCREEN-10 is a global patient-reported outcome (PRO) measure of well-being and health-related quality of life in children and adolescents aged 8-18 years. It includes 10 items that measure the subjective health and psychological, mental and social well-being experiences of children and adolescents over the past week. The scores for the 10 items are summed to produce a total score. This total score can then be transformed into a T-score or percentile rank, based on normative data, to facilitate interpretation. The higher the total score, the better the reported health-related quality of life (HRQoL).
Change from Baseline in Patient Global Impression of Severity (PGI-S) Depressive Symptoms at 24 Hours Post First Dose | Baseline (predose on Day 1) and 24 hours post first dose (i.e., Day 2)
  The PGI-S is a single PRO item that captures one's perceptions of the severity of his/her depressive symptoms over the past 24 hours. Participants will be asked to rate their disease severity using the following 5-point scale: 1 = None, 2 = Mild, 3 = Moderate, 4 = Severe, and 5 = Very severe. Higher scores indicate greater disease severity.
Change from Baseline in Clinical Global Impression - Severity Scale (CGI-S) Depressive Symptoms at 24 Hours Post First Dose | Baseline (pre-dose on Day 1) and 24 hours post first dose (i.e., Day 2)
  The CGI-S provides an overall clinician-determined summary measure of the severity of the participant's illness that considers all available information, including knowledge of the participant's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the participant's ability to function. The CGI-S will be used to rate the overall severity of illness on a scale of 1 to 7. Considering total clinical experience with the depression population, a participant is assessed on severity of illness at the time of rating according to the following scale: 1=normal (not at all ill); 2=borderline ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients. Higher scores indicate greater severity.

CONTACTS AND LOCATIONS:
Locations (1):
- Peachford Hospital-Atlanta Behavioral Research, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency